CLINICAL TRIAL: NCT03359603
Title: Electro-acupuncture of Different Treatment Frequency in Knee Osteoarthritis: a Pilot Randomized Clinical Trial
Brief Title: Electro-acupuncture in Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ping Zhou (Other)
Responsible Party: Sponsor-Investigator, Ping Zhou, Postgraduate, Beijing Hospital of Traditional Chinese Medicine
Organization: Beijing Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017BL-076-01
Record Dates: First submitted 2017-11-16; First posted 2017-12-02 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-11

CONDITIONS: Knee Osteoarthritis
Keywords: Electro-acupuncture; Knee osteoarthritis; Treatment frequency
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): After recruiting, patients are assigned to the group by randomization,and then receive electro-acupuncture treatment. Patients in the group will receive EA 3 sessions per week for 8 weeks. The EA stimulation lasted for 30 minutes with a dilatational wave of 2/100 Hz and a current intensity depending on the patient's comfort level (preferably with skin around the acupoints shivering mildly without pain).
  Interventions: Device: Electro-acupuncture
- Group B (Experimental): After recruiting, patients are assigned to the group by randomization,and then receive electro-acupuncture treatment. Patients in the group will receive EA once per week for 8 weeks. The EA stimulation lasted for 30 minutes with a dilatational wave of 2/100 Hz and a current intensity depending on the patient's comfort level (preferably with skin around the acupoints shivering mildly without pain).
  Interventions: Device: Electro-acupuncture

INTERVENTIONS:
Device: Electro-acupuncture — Patients will be treated by use of 5 obligatory and 3 customized acupoints. Obligatory points (ST35, EX-LE5, LR8, GB33 and Ashi) will be used in all patients. Other 3 customized acupoints should be chosen by the physicians on the basis of traditional Chinese medicine diagnosis for acupuncture channels related to the individual pain area, with the intent of optimizing efficacy. ST34, ST36, ST32, ST40 and EX-LE2 will be used for pain at stomach meridian. GB31, GB36, GB34, GB39 and GB41 will be used for pain at gallbladder meridian. BL39, BL40, BL57 and BL60 will be used for pain at bladder meridian. LR7, SP9, SP10, KI10, SP4, SP6, LR3 and KI3 will be used for pain at three yin meridians of foot. Needles will be stimulated manually for 10 seconds to achieve"De Qi". Paired alligator clips will be attached transversely to the needle holders at LR8-GB33 and two other customized acupoints. Other needles will be manipulated for 10 seconds during the treatments.

SUMMARY:
Knee osteoarthritis (KOA) is one of the most common musculoskeletal diseases in clinic. It usually occurs in middle-aged people, especially women. An estimated lifetime risk for KOA is approximately 40% in men and 47% in women. KOA is a chronic disease which can lead to obvious pain, joint stiffness, limitation of activity and even disability, with significant associated costs and effects on society, health systems, and individuals. The use of acupuncture as an approach for the management of chronic pain, is receiving increasing recognition from both the public and professionals. However, there are no universally accepted treatment frequency criteria in previous studies. The number of acupuncture treatments is no more than twice per week in most previous studies, while it is usually 3-5 sessions per week in clinical practice in China. The aim of this study is to compare the effects of different EA sessions (3 sessions per week versus once per week) in a pilot randomized controlled trial of KOA.

DETAILED DESCRIPTION:
Patients will be randomly allocated to one of two groups. In the 24-session treatments group (group A), patients will receive EA 3 sessions per week for 8 weeks. The EA stimulation lasted for 30 minutes with a dilatational wave of 2/100 Hz and a current intensity depending on the participant's comfort level (preferably with skin around the acupoints shivering mildly without pain). It involves having needles inserted into acupoints which are stimulated manually for 10 seconds to create "De Qi" sensation and paired alligator clips will be attached to the needle holders at LR8-GB33 and two other customized acupoints. Disposable needles (Huatuo) and the HANS-200A acupoint nerve stimulator (Nanjing Jisheng Medical Co., Ltd. production) will be used.

Patients in the 8-session treatments group (group B) will receive EA once per week for 8 weeks. Other interventions are the same as group A. Assessments will be conducted at baseline and 4, 6, 8, 12 and 16 weeks after randomization.

It is expected that the interventions will alleviate the sufferings of the patient. The risks of participation are minimal. Occasionally, acupuncture can make people feel nauseous or experience a temporary increase in pain either during or after treatment. Rare side effects during acupuncture treatment include fainting, infection and subcutaneous hematoma (pooling of blood under the skin). Participants will be warned of these potential side-effects before consenting to have acupuncture.

Patients will be allowed, or required, to back out of the trial based on the following:

1. A major protocol violation;
2. Development of a serious disease;
3. Adverse events related to electro-acupuncture;
4. Request to be back out of the trial. The purpose of the study is to accumulate clinical data, obtain the outcome data of the intervention method and prove the feasibility of the study protocol.

Sixty patients will be selected as the sample size according to clinical experience.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45-75 years old, male or female;
2. Single / bilateral knee pain, duration of more than 6 months;
3. KL (Kellgren-Lawrence) grade Ⅱ or Ⅲ in recent 6 months;
4. NRS ≥ 40mm;
5. Signed informed consent

Exclusion Criteria:

1. Surgery history of knee or waiting for surgery (knee replacement or knee arthroscopy);
2. Knee pain caused by other diseases (such as joint bodies, severe effusion of joint cavity, infection, malignant tumors, autoimmune diseases, trauma, etc.);
3. History of arthroscopy within 1 year or intra-articular injection within 4 months;
4. History of receiving acupuncture treatment within 3 months;
5. Severe acute/chronic organic or mental diseases;
6. Pregnant women, pregnant and lactating women;
7. Coagulation disorders (such as hemophilia, etc.);
8. Participation in another clinical study in the past 3 months;
9. With a cardiac pacemaker, metal allergy or needle phobia.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-12-25 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Response rate | baseline and 8 weeks
  the percentage of patients with improvement in average pain (numerical rating scale, NRS) at least 2 units and in Western Ontario and Mcmaster Universities Osteoarthritis Index (WOMAC) function subscale score at least 6 units at 8 weeks. Pain NRS was a self-administered instrument, a number selected from 0-10 by participant. Intensity of pain range (over past week): 0 =no pain to 10 =worst possible pain. Higher score indicating severe pain. The WOMAC function subscale referred to the participant's ability to move around and perform usual activities of daily living. The WOMAC function subscale was comprised of 17 questions regarding the degree of difficulty experienced due to OA in the study knee. The WOMAC function subscale score for each question ranged from 0 (minimum) to 4 (maximum), higher scores signified worse physical function. An overall score range of 0 (minimum) to 68 (maximum), with higher scores indicating worse physical function.

SECONDARY OUTCOMES:
Pain | baseline, 8 weeks and 16 weeks
  using numerical rating scale (NRS) and WOMAC pain subscale. Pain NRS was a self-administered instrument, a number selected from 0-10 by participant. Intensity of pain range (over past week): 0 =no pain to 10 =worst possible pain. Higher score indicating severe pain. The WOMAC pain subscale referred to the patient's pain. It was comprised of 5 items, with each item scored from 0 (minimum) to 4 (maximum), where 4 indicated worst pain condition. An overall score range of 0 (minimum) to 20 (maximum), with higher scores indicating worse physical function.
Knee-joint function | baseline, 8 weeks and 16 weeks
  using WOMAC function subscale. The WOMAC function subscale referred to the participant's ability to move around and perform usual activities of daily living. The WOMAC function subscale was comprised of 17 questions regarding the degree of difficulty experienced due to OA in the study knee. The WOMAC function subscale score for each question ranged from 0 (minimum) to 4 (maximum), higher scores signified worse physical function. An overall score range of 0 (minimum) to 68 (maximum), with higher scores indicating worse physical function.
Stiffness | baseline, 8 weeks and 16 weeks
  using WOMAC stiffness subscale. The WOMAC stiffness subscale was comprised of 2 questions regarding the degree of stiffness experienced in the study knee. The WOMAC stiffness subscale score for each question ranged from 0 (minimum) to 4 (maximum), higher scores signified worse stiffness. An overall score range of 0 (minimum) to 8 (maximum), with higher scores indicating more stiffness.
Overall effect | baseline, 8 weeks and 16 weeks
  using the Overall Treatment Effect (OTE)
Quality of life | baseline, 8 weeks and 16 weeks
  using the 12-Item Short Form Health Survey (SF-12)
Adverse events | up to 16 weeks
  using Adverse Event Form
Credibility score | 1 week（after the first treatment）
  using Credibility/expectancy questionnaire
Expectancy score | 1 week（after the first treatment）
  using Credibility/expectancy questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Cun-Zhi Liu, MD, Study Director — Beijing Hospital of Traditional Chinese Medicine
Locations (1):
- Beijing Hostipal of Traditional Chinese Medicine affiliated to Capital medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lin LL, Tu JF, Shao JK, Zou X, Wang TQ, Wang LQ, Yang JW, Sun N, Liu CZ. Acupuncture of different treatment frequency in knee osteoarthritis: a protocol for a pilot randomized clinical trial. Trials. 2019 Jul 11;20(1):423. doi: 10.1186/s13063-019-3528-8. PMID 31296249